CLINICAL TRIAL: NCT07287852
Title: Is Cerebonin (Egb761) a Disease-modifying Therapy in Mild Cognitive Impairment
Brief Title: A Pilot Study to Examine the Effect of Egb761 on Plasma Biomarker Levels and on Cognitive Function in Patients With MCI
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0658-22-HMO
Record Dates: First submitted 2025-06-29; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease (AD); Mild Cognitive Impairment (MCI)
Keywords: mild cognitive impairment; phosphorylated Tau; ginkgo biloba
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Ginkgo biloba extract

STUDY DESIGN:
Intervention Model Description: In this trial, all participants will be treated with Egb761. The investigators will evaluate plasma levels of phosphorylated Tau, cognitive performance and degree of behavioral impairment before treatment, and after 3 and 6 months of treatment. The change between pre-treatment plasma level of phosphorylated Tau versus post-treatment level, as well as change in cognitive and behavioral evaluations will be analyzed in each participant, to determine whether Egb761 induces an improvement in phosphorylated Tau level and whether it causes symptomatic relief.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A single arm trial, where all participants will receive the studied medication (Experimental): In this single arm trial, the post-treatment biomarkers levels will be compared to pre-treatment levels per participant, with each participant's pre-treatment biomarkers' levels serving as baseline for reference.
  Interventions: Dietary Supplement: Ginkgo Biloba Extract 761

INTERVENTIONS:
Dietary Supplement: Ginkgo Biloba Extract 761 — Each participant will receive two 120mg Egb761 pills per day along the 6 month trial

SUMMARY:
The goal of this clinical trial is to learn if the drug Egb761, produced from Ginkgo Biloba extract, works to improve the blood level of a biomarker of Alzheimer's disease, called phosphorylated-tau217 (p-tau217), which serves as a biomarker for disease activity in the brain. The main questions it aims to answer are:

Does drug Egb761 lower the plasma level of p-tau217 in patients with mild cognitive impairment? Does drug Egb761 improve cognitive and behavioral functions in these patients? Does Egb761 affect the blood levels of neurofilament-light (Nfl) and glial-fibrillary-acidic-protein (GFAP), which serve as additional biomarkers for brain disease activity?

Participants will:

Take Egb761 twice daily for 6 months Visit the clinic once every 3 months for checkups and tests Keep a diary of their symptoms

DETAILED DESCRIPTION:
Participating center: A single-center trial performed at Hadassah - Hebrew University Medical Center in Jerusalem, Israel. The investigators have vast experience in performing full medical and neuropsychological evaluations, and in performing clinical trials in patients with cognitive decline. Patients will be recruited via the cognitive Neurology clinics at the Hadassah Ein-Kerem campus, Hadassah Mount Scopus campus, and Merhav out-patient clinic for cognitive Neurology, which is associated and operated by Hadassah Neurologists.

Patient recruitment: 50 patients with mild cognitive impairment (MCI) will be recruited, according to its accepted definition. Patients with MCI will undergo standard evaluation, including brain imaging (MRI / CT), thyroid function tests, Vitamin B12, erythrocyte sedimentation rate (ESR), C-reactive protein (CRP) to rule out other causes of cognitive decline.

The investigators expect that approximately 70% of recruited patients will display increased plasma p-tau217 level, indicating MCI of Alzheimer's type.

Clinical and neuropsychological evaluation will include: (1) Full demographic data (age, gender, education level and occupation, family status, ethnicity and country of origin); (2) Clinical data on risk factors (metabolic/ cardiovascular risk factors - heart disease, diabetes, hypertension, hyperlipidemia; Infectious/ inflammatory risk factors - periodontal disease, systemic infections, systemic inflammatory conditions; Lifestyle factors - smoking, alcohol consumption, sleeping disorder, physical activity; and Mental factors - anxiety and depression, cognitive activity); (3) MoCA (in Hebrew version); (4) Mild Behavioral Impairment checklist (MBI-C), or Neuropsychiatric Inventory (NPI) questionnaire (in Hebrew version); (5) ADL and iADL questionnaire; (6)Trail making test -B (TMT-B); Word fluency test.

Determination of blood biomarkers: Venous blood will be drawn upon recruitment in a tube containing EDTA to prevent clotting. The blood will be centrifuged at 1200 rpm for 5 minutes, and plasma stored in -80°C, within two hours of drawing the blood sample. The samples will be stored in a temperature-controlled and monitored freezer, until delivery in dry ice to the central lab (Prof. Ben-Hur's lab at the Ein-Kerem campus) for determination of biomarkers. Blood samples that were collected at recruitment will be tested for p-tau217 level, neurofilament light and GFAP. The baseline p-tau217 will serve as a reference value for monitoring individual response to therapy, as well as the group trend in the other biomarkers.

Treatment: All patients will receive Cerebonin (Egb761) 240mg per day, by tablets of 120mg, taken twice daily.

Follow-up: After initiation of treatment, patients will be invited for follow-up visits at 3 months and 6 months. Clinical data (risk factor assessment), MoCA, MBI-C, iADL and plasma p-tau217 level will be evaluated in each visit. The investigators will evaluate total MoCA score, as well as its breakdown into cognitive domains (attention, executive, memory (both free and cued / recognition recall), visuospatial, language, and orientation). One point is added if the subject has ≤12 years of education.

Evaluating response to therapy: (1) In patients with high baseline plasma p-tau181 level, the investigators will compare pre- and post-treatment plasma p-tau-217 levels (Δp-tau). Since plasma p-tau217 is considered a biomarker of active brain disease, a reduction in its level will suggest a disease-modifying therapeutic effect; (2) The investigators will examine the trend in group averages of neurofilament and GFAP, as additional disease biomarkers. (3) The investigators will determine the symptomatic clinical response according to improvement in MoCA, MBI-C/NPI, TMT-B and ADL/iADL scores after 3 and 6 months of treatment; (4) The investigators will compare the treatment effect in MCI patients with high- versus normal- plasma p-tau217 levels (eg. in MCI of AD type versus non-AD type); (5) The investigators will examine the association between clinical improvement and change in the plasma level of biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Mild cognitive impairment, as defined by MoCA score of 19-25.
* Preserved instrumental activities of daily life (iADL).
* Clinical impression of MCI of AD type, and lack of major medical and neurological conditions, as detailed in the exclusion criteria.

Exclusion Criteria:

* Extrapyramidal signs, existence of multi-infract dementia, or Fronto-Temporal dementia, according to clinical impression by treating cognitive Neurologist.
* Active cancer, severe cardio-pulmonary disease or other medical condition which negatively affects ability to evaluate patients and complete follow-up.
* Inability to sign an informed consent due to psychiatric or dementing condition.
* Hypersensitivity to any ingredient of the study medication.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in plasma phosphorylated-tau level | Plasma biomarker level tested at recruitment, at 3 and 6-months of trial
  Change in post-treatment plasma phosphorylated Tau level (6 months time point) as compared to pre-treatment level. P-tau level is reported in pg/ml

SECONDARY OUTCOMES:
Symptomatic effect | The test will be performed at recruitment, at 3- and 6-months of treatment
  Change between pre-treatment and post-treatment (6 months time point) MoCA scores. MoCA score range is between 0-30.
Symptomatic effect | The test will be performed at recruitment, at 3- and 6-months of treatment
  Change between pre-treatment and post-treatment (6months time point) in TMT-B scores. TMT-B is measured as time (number of seconds) to complete the task.
Symptomatic effect | The test will be performed at recruitment, at 3- and 6-months of treatment
  Change between pre-treatment and post-treatment (6months time point) in word fluency score. Word fluency score is the number of words generated in the 1-minute timed test.
Symptomatic effect | The test will be performed at recruitment, at 3- and 6-months of treatment
  Change between pre-treatment and post-treatment (6 months time point) in the neuropsychiatric questionnaire score. The MBI-C questionnaire score range is 0-102.
Change in plasma GFAP level | Plasma biomarker will be determined at recruitment and at 3- and 6-months
  Change in post-treatment plasma GFAP level (6 months time point) as compared to pre-treatment level. GFAP level is reported in pg/ml.
Change in plasma neurofilament-light level | Plasma biomarker will be determined at recruitment and at 3- and 6-months
  Change in post-treatment plasma neurofilament-light level (6 months time point) as compared to pre-treatment level. Nfl level is reported in pg/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share IPD on cognitive, behavioral, and biomarker data without personal identification, as required by the IRB upon completion of the trial.